CLINICAL TRIAL: NCT06897189
Title: Optimizing Radiation Dose and Utilizing Wearable Devices to Reduce Arrhythmia Risk in Patients Undergoing Thoracic Radiotherapy: A Prospective Cohort Study
Status: Not yet recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2024-1631
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Cardiotoxicity; Thoracic Radiotherapy; Wearable Electronic Devices; Thoracic Neoplasms; Atrial Fibrillation
MeSH Terms: conditions — Cardiotoxicity; Thoracic Neoplasms; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective observational cohort study aims to assess the risk of radiation-induced cardiotoxicity in patients undergoing thoracic radiotherapy by integrating real-time arrhythmia monitoring using wearable cardiac rehabilitation (wearable CR) devices and AI-based cardiac substructure segmentation. The study will analyze radiation dose exposure to key cardiac structures, including the sinoatrial node (SAN) and pulmonary veins (PV), to identify risk factors for atrial fibrillation (AF) and other arrhythmias. Patients will receive wearable CR monitoring at 3, 12, and 24 months post-radiotherapy, with cardiology follow-up and intervention based on standard clinical guidelines. The study will recruit 111 patients over three years, with a two-year follow-up after radiotherapy. The primary endpoint is the incidence of grade 3+ AF within 2 years, with secondary outcomes including any-grade arrhythmia rates, arrhythmia burden, and survival analysis. By establishing a prospective thoracic radiotherapy patient cohort, this study aims to identify dose-related risk factors, improve early detection and management of radiation-induced arrhythmias, and provide evidence-based strategies to enhance treatment safety and efficacy.

DETAILED DESCRIPTION:
"This prospective observational cohort study aims to assess the risk of radiation-induced arrhythmias in patients undergoing thoracic radiotherapy for solid tumors, integrating real-time cardiac monitoring with wearable cardiac rhythm (Wearable CR) devices and AI-based cardiac substructure segmentation. The study will recruit 111 patients over three years, with a two-year follow-up post-radiotherapy. Patients will undergo Wearable CR monitoring at 3, 12, and 24 months, facilitating early detection and intervention based on standard cardiology guidelines. Radiation dose exposure to key cardiac structures, including the sinoatrial node (SAN) and pulmonary veins (PV), will be analyzed to evaluate correlations with atrial fibrillation (AF) and other arrhythmias. AI-driven segmentation will aid in optimizing dose distribution to minimize cardiotoxicity while maintaining treatment efficacy. The primary endpoint is the incidence of grade 3+ AF within 2 years, with secondary endpoints including any-grade arrhythmia rates, arrhythmia burden, and survival outcomes. All enrolled patients will receive standard radiotherapy protocols tailored to their respective cancer types, ensuring treatment consistency while assessing the impact of radiation on any kinds of cardiotoxicities.

ELIGIBILITY:
Inclusion Criteria:

* Patients with solid tumors requiring thoracic radiotherapy
* Undergoing curative-intent radiotherapy
* Expected survival > 4 months
* Adults aged ≥ 20 years
* ECOG performance status 0-2
* Classified as moderate-to-high risk for radiation-induced cardiotoxicity per the 2022 ESC guidelines
* Able to read, understand, and sign the informed consent form

Exclusion Criteria:

* History of prior thoracic radiotherapy
* Inability to provide informed consent or refusal to participate
* Pre-existing arrhythmia diagnosed through medical history or pre-treatment evaluation
* Expected survival ≤ 4 months
* Classified as low risk for radiation-induced cardiotoxicity per the 2022 ESC guidelines
* Unsuitability for Wearable CR device use

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing thoracic radiotherapy for solid tumors with curative intent, aged ≥ 20 years, ECOG 0-2, and at moderate-to-high risk for radiation-induced cardiotoxicity per ESC 2022 guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 111 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2030-02-16 (Estimated); Study Completion 2030-02-16 (Estimated)

PRIMARY OUTCOMES:
Incidence of Grade 3 or Higher Atrial Fibrillation (AF) within 2 Years After Radiotherapy | Up to 2 years post-radiotherapy
  The proportion of patients who develop Grade 3 or higher atrial fibrillation within 2 years following thoracic radiotherapy.

SECONDARY OUTCOMES:
Incidence of Any-Grade Atrial Fibrillation (AF) within 2 Years After Radiotherapy | p to 2 years post-radiotherapy
  The proportion of patients experiencing any grade of atrial fibrillation within 2 years of radiotherapy.
Incidence of Any-Grade Arrhythmia within 2 Years After Radiotherapy | Up to 2 years post-radiotherapy
  The proportion of patients who develop any type of arrhythmia within 2 years of radiotherapy.
ypes and Frequency of Arrhythmias Occurring Within 2 Years After Radiotherapy | Up to 2 years post-radiotherapy
  Classification and frequency analysis of different types of arrhythmias detected within 2 years after radiotherapy.
Incidence of Any-Grade Arrhythmia within 3 Months After Radiotherapy | Up to 3 months post-radiotherapy
  The proportion of patients who develop any-grade arrhythmia within 3 months after radiotherapy.
Incidence of Any-Grade Arrhythmia within 1 Year After Radiotherapy | Up to 1 year post-radiotherapy
  The proportion of patients experiencing any-grade arrhythmia within 1 year of radiotherapy.
Overall Survival (OS), Cancer-Specific Survival (CSS), and Progression-Free Survival (PFS) | Up to 2 years post-radiotherapy
  Time from radiotherapy to death from any cause, CSS: Time from radiotherapy to death due to cancer, PFS: Time from radiotherapy to disease progression or death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei Cancer Center, Yonsei University College of Medicine, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No